CLINICAL TRIAL: NCT05823129
Title: Effectiveness of Telerehabilitation on Quality of Life and Mobility of Early Post-discharge Hip Fracture Patients
Brief Title: 'Home Sweet Home' Programme-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 22-095
Record Dates: First submitted 2022-10-27; First posted 2023-04-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Geriatric Hip Fracture
Keywords: Empowerment; Telerehabilitation; Geriatric Hip Fractures; Functional outcomes
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A project manager will randomize the participants to the intervention or standard-care group, and the outcome assessor will not be informed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (No Intervention): Usual clinical protocol is followed, the caregiver is given verbal training and assistive instructions by therapists and clinicians before patient discharge. Brief pamphlets are provided on post-operative care of patients. Patients are encouraged to perform rehabilitative exercises according to "what they have learned" during the in-patient stay.
  "Remote-TUG" app is only used in the first and final assessment at day 30.
- Intervention Group (Experimental): A recruitment assessment videoconference is scheduled at the 1st post-discharge week providing clear instructions on how to perform daily TUG test. The TUG test is to be performed at least twice in the morning and twice afternoon and complimented by other specific training exercises as specified in HSH1. Training instructions and assessment is performed by videoconference to ascertain that both the patient and the caregiver can follow instructions in using the "remote-TUG" smartphone app and safety measures are understood and applied when assisting the patients in exercises. Clear video instructions and multimedia for review will be provided. Interim videoconference will be conducted again after week 2 to ascertain adherence. Non-adherence can be immediately detected by remote data collection from the "remote-TUG" server interface. Non-adherence will trigger phone calls and videoconferences serving as reminders and performing troubleshooting.
  Interventions: Behavioral: Tele-rehabilitation caregiver empowerment enhanced post- discharge rehabilitation directive

INTERVENTIONS:
Behavioral: Tele-rehabilitation caregiver empowerment enhanced post- discharge rehabilitation directive — The intervention group will receive an implemented TUG test-based telerehabilitation program. The TUG test-based telerehabilitation involves patients routinely doing two TUG tests by themselves twice daily. Each patient will be provided with a unique link to the TUGstopwatch, a prerecorded video outlining instructions on how to properly conduct a TUG test, and support and guidance for patients and caregivers throughout the study period.
  Arms: Intervention Group

SUMMARY:
Objectives:

To determine the effectiveness of telerehabilitation on the quality of life and mobility of early post-discharge in hip fracture patients, and to investigate whether telerehabilitation in the form of daily TUG tests recorded digitally will improve recovery outcomes for post-surgery hip fracture patients.

Hypothesis to be tested:

Main hypothesis: Caregiver empowerment can improve functional walking and quality of life at 1 month after discharge Secondary hypothesis: Hospital readmission and mortality rate can be reduced.

Design and subjects:

This is a prospective randomised controlled trial and subjects are fracture hip patients

Instruments:

Timed-Up-and-Go (TUG) test, EuroQol EQ5D-5L, Parker Mobility score

Interventions:

A videoconference scheduled at the 1st post-discharge week provides clear instructions and directions on how to perform daily exercise prescriptions based on the TUG test. Video instructions and multimedia for review will be provided. Interim videoconference will be conducted again after week 2 to ascertain adherence.

Main outcome measures:

Primary outcomes:

Timed-Up-and-Go (TUG) test taken at day 0 and 28

Secondary outcome:

EQ5D-3L and Parker Mobility Score taken on day 0 and 28

Other covariates Patient baseline demographics Classification of hip fractures Type of surgical intervention Comorbidities

Any adverse events occurring:

* Severe adverse events including: unplanned hospital readmissions, fall injury causing fractures, failure of internal fixation, death
* Other adverse events including: unplanned clinic visits, complications requiring change in rehabilitation plan or additional medical/ surgical intervention, complications requiring closer observation

Data analysis:

Shapiro-Wilk test and independent sample t-test is performed for variables to ascertain normal distribution and compared for main outcomes. Binary variables and categorical variables with Chi-squared tests. Time-based outcomes are compared using Kaplan-Meier time to event analysis and log-rank test. A type 1 error rate / p value of 0.05 is used for statistical significance.

Expected results:

Fracture hip patients can be benefited from the empowerment program

DETAILED DESCRIPTION:
Rehabilitation after hip fracture surgery is crucial in the recovery process for hip fracture patients. Although huge emphasis has been placed on the importance of undertaking post-surgery daily exercise routines to patients, some patients still neglect these exercise routines due to various reasons, leading to insufficient recovery.

The Geriatric Hip Fracture Clinical Pathway (GHFCP) is first designed and implemented in the Hong Kong West Cluster. The implementation of the GHFCP resulted in a decreased preoperative and total length of stay, decreased surgical site infection, decreased pressure sore, decreased 30-days and 12-months mortality rate.

GHFCP specifically streamline acute and rehabilitation in-patient healthcare delivery and ends after the patient is discharged.

Through many studies, telerehabilitation has proven to promote recovery in post-surgery patients, especially those that had undergone orthopaedic surgery. Present evidence indicates a strong positive effect for patients undergoing telerehabilitation post-orthoepaedic surgery, with a systematic review and meta-analysis suggesting that "increased intensity provided by telerehabilitation is a promising option to be offered to patients."

At the same time, the Timed-up-and-Go (TUG) test has proven to be an accurate and objective assessment of the physical mobility of geriatric individuals. It is quick and easy to perform without the requirement for special equipment or training. When utilized as a descriptive tool, Timed-up-and-Go test data can detail a patient's balance, gait speed, and functional ability. As such, it is a suitable test to be utilized for telerehabilitation due to its easy operation and ability to communicate sufficient patient data, all of which can be done in a patient's own home and sent electronically through the internet to healthcare professionals. TUG when performs daily may incent by patients' adherence to rehabilitation in form of a biofeedback loop.

With evidence displaying the effectiveness of the TUG test and telerehabilitation in their respective fields, this research aims to combine the two and provide telerehabilitation in the format of regular TUG tests in conjunction with an e-response system, encouraging patients to perform the exercise appropriately, thus improving their post-surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have provided informed consent to be included in the study
* Geriatrics ≥ 65 years of age
* Suffered hip fracture accompanied by successful surgery

  * Less than 2 weeks following patient discharge from rehabilitation
  * Less than four months post-operation
* Patients capable of walking on fracture without endangering their fracture fixation,
* Patients have been taught how to walk in the rehabilitation centre
* Caretaker/family has the ability to conduct the TUG test

  * patient's residence is spacious enough to safely perform TUG test
  * Video calling showing the performance of the TUG test should be supported
  * Caretaker should have basic technological competency
  * Caretaker should have sufficient cognitive ability to understand the TUG test
  * Caretaker should have the ability to supervise patient during the TUG test
* Patients should have similar post-surgery recovery progress

  * Record at the start if each patient requires assistance - with or without aid, e.g. walking frame etc
  * Should at least have the potential to walk

Exclusion Criteria:

* Patients with multiple fractures affecting mobility
* chair-bound or bed-bound
* Patients with severe cognitive impairment

  * Assessed based on:

    * unable to follow command to walk
    * unable to identify time, person and space
* Presence of terminal illnesses/diseases
* Presence of multiple medical illnesses

  * Determined by the Charleson comorbidity score

    * Patients excluded if the score is larger or equal to 6

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-07-16 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in Walking function between Day 0 and Day 28 | Change in TUG test between Day 0 and Day 28
  Timed-Up-and-Go (TUG) test

SECONDARY OUTCOMES:
Change in Health-related quality of life between Day 0 and Day 28 | Change in quality of life between Day 0 and Day 28
  The EQ5D-5L is a patient-reported outcome measure of health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is rated on scale that describes the degree of problems in that area. This tool also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable.
Change in Patient's mobility measured by Parker Mobility Score between Day 0 and Day 28 | Change in mobility score between Day 0 and Day 28
  The Parker Mobility Score is a composite measurement of the patient's mobility indoors, outdoors, and during shopping. It is a 3-item patient-reported measure, each item valued 0-3 points, the total score ranges from 0 (worst possible mobility) to 9 (best possible mobility)
Incidence of severe adverse events | Day 28
  Incidence of unplanned hospital readmissions, fall injury causing fractures, failure of internal fixation, death will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong